CLINICAL TRIAL: NCT05464914
Title: Post Extraction Wound Healing Evaluation of Immediate Complete Denture Using IPR Scale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Shady El Naggar, Clinical Professor, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01154777474
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Complete Edentulism Due to Periodontal Disease (Disorder)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional upper immediate denture (No Intervention): Conventional upper immediate denture without any surgical lining
- Upper immediate denture lined by surgical dressing (Active Comparator): Upper immediate denture lined by surgical dressing using CEO Pack dressing
  Interventions: Drug: CEO Pack

INTERVENTIONS:
Drug: CEO Pack — is a eugenol-free, surgical dressing and periodontal pack that has no burning sensation, no unpleasant taste or odor, and offers proven protection to surgical sites. This product promotes cleanliness and healing. Plastic and cohesive, ropes of any length or thickness can be formed. The smooth texture allows this product to adapt closely to the teeth and tissue in order to protect the wound. It sets with resilient, non-brittle hardness.
  Other Names: Perio pak; Surgical pak
  Arms: Upper immediate denture lined by surgical dressing

SUMMARY:
In the first part, after a brief introduction, the advantages and disadvantages of immediate dentures are compared. There is a detailed discussion on assessment and treatment planning which includes history taking, examination of the soft and hard tissues, current prostheses, occlusion as well as discussion on investigations required and formulating a diagnosis. The first part ends with a summary of types of immediate dentures and denture designs.

DETAILED DESCRIPTION:
An Immediate denture is a complete or partial removable prosthesis that is fitted immediately after extraction or modification of teeth. The prosthesis replaces the missing/modified teeth and where required, the adjacent hard and soft tissues. It is constructed prior to the extraction of teeth and is used immediately to provide function and aesthetics which are lost as a result of tooth removal and avoid the embarrassment patients may have with living without teeth, while waiting for the tissues to heal prior to definitive tooth replacement.1 (See image 1) Some clinicians take impressions on the day of the extractions and fit the dentures a few days later. These dentures are fraught with challenges as the alveolar ridge begins to resorb soon after. Therefore an immediate denture is only truly an immediate denture when fitted on the day of the extractions.

The use of a removable prosthesis within the UK is currently around 19% of adults in the general population 2 and in spite of this decreasing trend, as patients retain their natural dentition into older age,2 there is still a need for prosthodontic replacement as teeth are lost as a result of caries, periodontal disease, tooth wear or trauma. 3,4,5 The provision of an immediate denture can be challenging and close co-operation between patient, technician, and clinician is required.

ELIGIBILITY:
Inclusion Criteria:

* Good physical and mental health
* Willing to give informed consent
* Normal maxilla-mandibular relationship Angle Class I
* Adequate bone quality and quantity in terms of width and height in the anterior maxillary and mandibular ridges verified by preoperative cone beam CT
* Adequate inter-arch space to accommodate maxillary and mandibular implant prostheses

Exclusion Criteria:

* Uncontrolled diabetes
* Smoking habits
* Radiotherapy
* Clinical or radiographic signs of pathologic conditions, osteoporosis
* Patients on corticosteroids
* Bruxism

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Post extraction Assessment | 6 weeks
  Post extraction Assessment of Wound Healing following Inflammatory Proliferative Remodeling (IPR) scale. The scale is divided into three subscales corresponding to the three phases of wound healing, and each is rated at the appropriate time point during follow-up,3 yielding three subscale scores and a total score. The outcome parameters of the subscales depend on the biological events that occur during that specific phase. At the end of follow up, the total score of the IPR Scale was calculated (0-16), where 0-4 indicated poor healing, 5-10 acceptable healing, and 11-16 excellent healing

CONTACTS AND LOCATIONS:
Overall Officials: Shady M. El Naggar, PhD, Principal Investigator — Badr University in Cairo
Locations (1):
- Shady Elnaggar, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT05464914/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT05464914/SAP_003.pdf
  • Informed Consent Form (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT05464914/ICF_004.pdf